

Version Date: 09/20/2021

TO: ALL NATIONAL CANCER CLINICAL TRIALS NETWORK (NCTN) MEMBERS; CTSU

FROM: , Protocol Coordinator II (E-mail:

RE: <u>\$1605</u>, "Phase II Trial of Atezolizumab in BCG-Unresponsive Non-Muscle Invasive

Bladder Cancer." Study Chairs: Drs. P. Black, P. Singh, and S. Lerner.

**REVISION #9** 

Study Chair: Peter C.V. Black, M.D. Phone number: 605/875-4301 E-mail: pblack@mail.ubc.ca

Action Codes

(√) Expedited review allowed

**Key Updates** 

(√) Data Submission / Forms changes
 (√) Editorial / Administrative changes

**Sites using the CIRB as their IRB of record:** The protocol and/or informed consent form changes have been approved by the CIRB and must be activated within 30 days of the CIRB posting of this notice.

Sites not using the NCI CIRB: Per CTMB Guidelines, the protocol updates and/or informed consent changes must be approved by local IRBs within 90 days of distribution of this notice.

#### **REVISION #9**

This revision has been prepared to add forms and data collection elements from Genentech.

#### Protocol Changes

- The version date has been updated.
- Section 14.4k: A sentence has been added to note to Submit documentation supporting findings of metastatic bladder cancer, muscle-invasive bladder cancer (e.g. pathology report).
- Section 14.4I: This section has been updated to note the instructions to submit pathology and operative reports from cystectomy procedures.
- Section 14.4p: This section has been added to note the forms to submit within 30 days after the distribution of revision #9.
- 5. <u>Section 14.4q:</u> This section has been added to note the electronic signature page to be submitted within 15 days after submission of all data requested in revision #9.
- Section 18.5: This section has been added to note the Investigator Electronic Signature instructions.

4201 Medical Drive, Suite 250 | San Antonio, TX 78229 | OFFICE 210-614-8808 | FAX 210-614-0006





#### **Model Consent Form Changes**

The version date has been updated.

The updated protocol and model consent form can be accessed from the CTSU website (<a href="www.ctsu.org">www.ctsu.org</a>). Please discard any previous versions of the documents and replace with the updated versions. Please contact <a href="mailto:ququestion@crab.org">ququestion@crab.org</a> or 206/652-2267 with any questions.

This study has been reviewed and approved by the NCI's Central Institutional Review Board (CIRB).

This memorandum serves to notify the NCI, and SWOG Statistics and Data Management Center.

cc: PROTOCOL & INFORMATION OFFICE

- Genentech

# Informed Consent Model for **S1605**

#### \*NOTES FOR LOCAL INSTITUTION INFORMED CONSENT AUTHORS:

This model informed consent form has been reviewed by the DCTD/NCI and is the official consent document for this study. Local IRB changes to this document are allowed. (Institutions should attempt to use sections of this document that are in bold type in their entirety.) Editorial changes to these sections may be made as long as they do not change information or intent. If the institutional IRB insists on making additions, deletions, or more substantive modifications to the risks or alternatives sections, they may be justified in writing by the investigator and approved by the IRB. Under these circumstances, the revised language, justification and a copy of the IRB minutes must be forwarded to the SWOG Operations Office for approval before a patient may be registered to this study.

Please particularly note that the questions related to banking of specimens for future study are in bolded type and may not be changed in any way without prior approval from the SWOG Operations Office.

| Readability Statistics: | | |
|----------------------------|------|----------------------|
| Flesch Reading Ease | 57.6 | (targeted above 55) |
| Flesch-Kincaid Grade Level | 9.4 | (targeted below 8.5) |

- Instructions and examples for informed consent authors are in [italics].
- A blank line, \_\_\_\_\_\_, indicates that the local investigator should provide the
  appropriate information before the document is reviewed with the prospective
  research participant.
- The term "study doctor" has been used throughout the model because the local investigator for a cancer treatment trial is a physician. If this model is used for a trial in which the local investigator is not a physician, another appropriate term should be used instead of "study doctor".
- The dates of protocol updates in the header and in the text of the consent is for reference to this model only and should not be included in the informed consent form given to the prospective research participant.
- The local informed consent must state which parties may inspect the research records. This includes the NCI, the drug manufacturer for investigational studies, any companies or grantors that are providing study support (these will be listed in the protocol's model informed consent form) and SWOG.

"SWOG" must be listed as one of the parties that may inspect the research records in all protocol consent forms for which patient registration is being credited to SWOG. This includes consent forms for studies where all patients are registered directly through the SWOG Data Operations Office, all intergroup studies for which the registration is being credited to SWOG (whether the registration is through the SWOG Data Operations Office or directly through the other group), as well as consent forms for studies where patients are registered via CTSU and the registration is credited to SWOG.



• When changes to the protocol require revision of the informed consent document, the IRB should have a system that identifies the revised consent document, in order to preclude continued use of the older version and to identify file copies. An appropriate method to identify the current version of the consent is for the IRB to stamp the final copy of the consent document with the approval date. The stamped consent document is then photocopied for use. Other systems of identifying the current version of the consent such as adding a version or approval date are allowed as long as it is possible to determine during an audit that the patient signed the most current version of the consent form.

#### \*NOTES FOR LOCAL INVESTIGATORS:

- The goal of the informed consent process is to provide people with sufficient information for making informed choices about participating in research. The consent form provides a summary of the study, the individual's rights as a study participant, and documents their willingness to participate. The consent form is, however, only one piece of an ongoing exchange of information between the investigator and study participant. For more information about informed consent, review the "Recommendations for the Development of Informed Consent Documents for Cancer Clinical Trials" prepared by the Comprehensive Working Group on Informed Consent in Cancer Clinical Trials for the National Cancer Institute. The Web site address for this document is <a href="http://cancer.gov/clinicaltrials/understanding/simplification-of-informed-consent-docs/">http://cancer.gov/clinicaltrials/understanding/simplification-of-informed-consent-docs/</a>
- Suggestion for Local Investigators: An NCI pamphlet explaining clinical trials is available for your patients. The pamphlet is titled: "Taking Part in Cancer Treatment Research Studies". This pamphlet may be ordered on the NCI Web site at <a href="https://cissecure.nci.nih.gov/ncipubs">https://cissecure.nci.nih.gov/ncipubs</a> or call 1-800-4- CANCER (1-800-422-6237) to request a free copy.
- Optional feature for Local Investigators: Reference and attach drug sheets, pharmaceutical information for the public, or other material on risks. Check with your local IRB regarding review of additional materials.



<sup>\*</sup>These notes for authors and investigators are instructional and should not be included in the informed consent form given to the prospective research participant.

# Study Title for Study Participants: Testing the use of Atezolizumab Immunotherapy in Non-Muscle Invasive Bladder Cancer that has Not Responded to Prior Bacillus Calmette-Guerin (BCG) Therapy

# Official Study Title for Internet Search on http://www.ClinicalTrials.gov: <u>S1605</u>, "Phase II Trial of Atezolizumab in BCG-Unresponsive Non-Muscle Invasive Bladder Cancer"

This is a clinical trial, a type of research study. Your study doctor will explain the clinical trial to you. Clinical trials include only people who choose to take part. Please take your time to make your decision about taking part. You may discuss your decision with your friends and family. You can also discuss it with your health care team. If you have any questions, you can ask your study doctor for more explanation.

## What is the usual approach to my non-muscle invasive bladder cancer?

You are being asked to take part in this study because you have superficial bladder cancer that has not invaded into the bladder muscle wall and that did not respond to Bacillus Calmette-Guerin (BCG). Unless the person is in a study, when people do not respond to BCG, or the FDA approved drug Valrubicin, or other treatments individualized to a person's clinical situation, treatment usually involves removal of the bladder (cystectomy). This study will test how effective the investigational immunotherapy drug atezolizumab is at keeping non-muscle invasive bladder cancer from coming back or getting worse. The study drug, atezolizumab, although approved by the FDA to treat other stages of bladder and lung cancers, is not approved by the FDA for treatment of bladder cancer at this early stage.

# What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- you may choose to have the usual approach described above without being in a study
- you may choose to take part in a different study, if one is available
- or you may choose not to be treated for cancer but you may want to receive comfort care to relieve symptoms

# Why is this study being done?

The purpose of this study is to test the good and bad effects of the investigational immunotherapy drug atezolizumab in stopping non-muscle invasive bladder cancer from coming back and progressing to muscle invasive bladder cancer. Atezolizumab is not approved by the FDA for treatment of this type of cancer. Atezolizumab is a type of immunotherapy (a drug that helps your body to fight a specific part of each cancer cell). About 202 people will take part in this study.



# What are the study groups?

All study participants will get the same study treatment. You will receive atezolizumab into a vein once every 21 days for up to 17 times. If your cancer stops responding, you will stop taking the study drug.

About 13 weeks after you start the study, you will have a test (cystoscopy) that allows the doctor to look at the lining of your bladder to see whether the cancer is responding to the treatment. After that you will have the cystoscopy again about every 3 months. Tissue samples of the lining of your bladder may also be taken during cystoscopy if it is suspected that the cancer has returned. If those samples also suggest that the cancer has returned, you will have a biopsy or TURBT.

If you have a type of bladder cancer called carcinoma in situ (CIS), you will probably have a biopsy about 25 weeks after you start the study. You will not need to have this biopsy if you had a negative biopsy at week 13.

## How long will I be in this study?

You will get the study drug once every 21 days for up to 17 times. If there are no treatment delays, you will take the study drug for about 1 year, or as long as your disease does not get worse and the side effects are not too severe. After you finish the study drug, your doctor will continue to watch you for side effects and follow your condition for up to five years.

# What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual
- You may be asked sensitive or private questions which you normally do not discuss

The atezolizumab used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the atezolizumab or the study approach.

Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.



Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

The tables below show the most common and the most serious side effects that researchers know about. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Risk Profile for Atezolizumab (CAEPR Version 2.2, July 23, 2018) (updated 9/10/18)

## COMMON, SOME MAY BE SERIOUS

In 100 people receiving atezolizumab (MPDL3280A), more than 20 and up to 100 may have:

- Tiredness
- Infection



#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving atezolizumab (MPDL3280A), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Diarrhea, nausea, vomiting
- Difficulty swallowing
- Fever
- Flu-like symptoms including body aches
- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness
  of breath, swelling of the face or throat
- · Reaction during or following a drug infusion which may cause fever, chills, rash
- Loss of appetite
- Pain in back
- Cough, shortness of breath, stuffy nose
- Itching, acne, rash

Atezolizumab (MPDL3280A) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Hormone gland problems (especially the thyroid, pituitary and adrenal glands, and pancreas). Signs and symptoms may include: headaches that will not go away or unusual headaches, extreme tiredness or changes in mood or behavior decreased sex drive; weight loss or weight gain; excessive thirst or urine; dizziness or fainting.
- Pain in belly
- Pain or swelling of the joints
- Rash that develops on skin, nails, scalp and inside of mouth or vagina that may be painful



#### RARE, AND SERIOUS

In 100 people receiving atezolizumab(MPDL3280A), 3 or fewer may have:

Bruising, bleeding

Atezolizumab (MPDL3280A) may cause your immune system to attack normal organs and cause side effects in many parts of the body. These problems may include but are not limited to:

- Heart problems including swelling and heart failure. Symptoms and signs of heart problems may include: shortness of breath, swelling of the ankles and body.
- A condition with high blood sugar which leads to tiredness, frequent urination or excessive thirst
- Swelling and redness of the eye
- Intestinal problems (colitis) that can rarely lead to tears or holes in your intestine.
   Signs and symptoms of colitis may include: diarrhea or increase in bowel movements, blood in your stools or dark, tarry, sticky stools, severe belly pain or tenderness.
- Liver problems (hepatitis) which can cause liver failure. Signs and symptoms of hepatitis may include: yellowing of your skin or the whites of your eyes, severe nausea or vomiting; drowsiness; pain in the right upper belly.
- Swelling of the brain (meningitis/encephalitis), which may cause: headache, confusion, sleepiness, seizures, and stiff neck
- Problem of the muscle, including swelling, which can cause muscle pain and severe muscle weakness sometimes with dark urine
- Problem of the nerves that can cause paralysis. Signs and symptoms may include: numbness, tingling of hands and feet; weakness of the arms, legs.
- Kidney problems, including nephritis and kidney failure requiring dialysis. Signs
  of kidney problems may include: decrease in the amount of urine, blood in your
  urine, ankle swelling.
- Lung problems (pneumonitis and pleural effusion). Symptoms may include: new or worsening cough, chest pain, shortness of breath.
- Skin: blisters on the skin

The CT scan that you will receive in this study will expose you to low amounts of radiation. Every day, people are naturally exposed to low levels of radiation that come from the sun and the environment. This type of radiation is called "background radiation". No one knows for sure whether exposure to low amounts of radiation is harmful for your body. However, scientists believe that being exposed to too much radiation can cause harmful side effects, including causing a new cancer.



Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

Reproductive risks: You should not get pregnant, breastfeed, or father a baby while in this study. The atezolizumab used in this study could be very damaging to an unborn baby.

Check with the study doctor about what types of birth control, or pregnancy prevention, to use. You must use birth control for 150 days after your last treatment with atezolizumab. If you or your partner becomes pregnant, contact the study doctor immediately.

# What possible benefits can I expect from taking part in this study?

Taking part in this study may or may not make your health better. The researchers hope that atezolizumab will be helpful, but we do not know that it will be. This study may help researchers learn things that may help other people in the future.

# Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- · If you do not follow the study rules
- If the study is stopped by the sponsor (SWOG), IRB or FDA. The IRB (Institutional Review Board) is a group of people who review the research with the goal of protecting the people who take part in the study

# What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

| For questions about your rights while in this study, call the | (insert |
|---|---|
| name of center) Institutional Review Board at | (insert telephone number). |
| (Note to Local Investigator: Contact information for patient | representatives or other individuals |
| at a local institution who are not on the IRB or research tea | m but take calls regarding clinical |
| trial questions can also be listed here.) | |



## What are the costs of taking part in this study?

The atezolizumab will be supplied at no charge while you take part in this study. The cost of getting the atezolizumab ready and giving it to you is not paid by the study sponsor so you or your insurance company may have to pay for this. It is possible that the atezolizumab may not continue to be supplied while you are on the study. Although it is not likely, if this happens, your study doctor will talk to you about your options.

You and/or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this study, including the cost of tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are supplied at no charge. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be charged for any testing that is done with your specimens.

You will not be paid for taking part in this study.

## What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.

# Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.



There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The study sponsor (SWOG) and the drug company supporting the study (Genentech).
- Your local Institutional Review Board, IRB, is a group of people who review the research
  with the goal of protecting the people who take part in the study.
- The Food and Drug Administration and the National Cancer Institute in the U.S., and similar ones if other countries are involved in the study.
- The Cancer Trials Support Unit (CTSU), a research group sponsored by the National Cancer Institute (NCI) to provide greater access to cancer trials.
- Alliance, NRG, and ECOG-ACRIN, research groups sponsored by the National Cancer Institute (NCI)

# Where can I get more information?

You may visit the NCI Web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

[Note to Informed Consent Authors: the above paragraph complies with the new FDA regulation found at 21CFR50.25 (c) and must be included verbatim in all informed consent documents. The text in this paragraph cannot be revised.]

# Who can answer my questions about this study?

| You can talk to the study doc | tor about any questions or concerns yo | ou have about this study or to |
|---|---|---|
| report side effects or injuries. | Contact the study doctor | (insert name of |
| study doctor[s]) at | (insert telephone number) | ). |



#### ADDITIONAL STUDIES SECTION:

## This section is about optional studies you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. You will not get health benefits from any of these studies. The researchers leading this optional study hope the results will help other people with cancer in the future.

The results will not be added to your medical records, and you or your study doctor will not know the results.

You will not be billed for these optional studies. You can still take part in the main study even if you say 'no' to any or all of these studies. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies.

## 1. Future Contact

I agree to allow my study doctor, or someone approved by my study doctor, to contact me regarding future research involving my participation in this study.

Yes No

# 2. Optional Biobanking for Possible Future Studies

Researchers are trying to learn more about cancer, diabetes, and other health problems. Much of this research is done using samples from your tissue, blood, urine, or other fluids. Through these studies, researchers hope to find new ways to prevent, detect, treat, or cure health problems.

Some of these studies may be about genes. Genes carry information about features that are found in you and in people who are related to you. Researchers are interested in the way that genes affect how your body responds to treatment.

If you choose to take part, tissue, blood, and urine will be collected. The researchers ask your permission to store and use your samples and related health information (for example, your response to cancer treatment, or results of study tests and medicines you are given) for medical research. The research that may be done is unknown at this time. Storing samples for future studies is called "biobanking". The Biobank is being run by SWOG and is supported by the National Cancer Institute.



#### WHAT IS INVOLVED?

If you agree to allow your specimens to be stored and used in future research, here is what will happen next:

- 1) A sample from the tissue that was collected at the time of your surgery will be sent to the Biobank. During the study if your doctor collects tissue to check to see if your disease is coming back, extra tissue will be collected. Also, a small amount of blood (one to two teaspoons) will be taken prior to beginning treatment during Weeks 1, 4, 7 and 13. Urine (about 2 Tablespoons) will be taken during Weeks 1, 13, 25, 49 and 73 of the study. If you agree below, all of these specimens will be saved for future research studies.
- 2) Your sample and some related health information may be stored in the Biobank, along with samples and information from other people who take part. The samples will be kept until they are used up. Information from your medical record will be updated from time to time.
- 3) Qualified researchers can submit a request to use the materials stored in the Biobanks. A science committee at the clinical trials organization, and/or the National Cancer Institute, will review each request. There will also be an ethics review to ensure that the request is necessary and proper. Researchers will not be given your name or any other information that could directly identify you.
- 4) Neither you nor your study doctor will be notified when research will be conducted or given reports or other information about any research that is done using your samples.
- 5) Some of your genetic and health information may be placed in central databases that may be public, along with information from many other people. Information that could directly identify you will not be included.

## WHAT ARE THE POSSIBLE RISKS?

- The most common risks related to drawing blood from your arm are brief pain and possibly a bruise.
- There is a risk that someone could get access to the personal information in your medical records or other information researchers have stored about you.
- 3) There is a risk that someone could trace the information in a central database back to you. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.
- 4) In some cases, genetic information could be used to make it harder for you to get or keep a job or insurance. There are laws against the misuse of genetic information, but they may not give full protection. There can also be a risk in knowing genetic information. New health information about inherited traits that might affect you or your blood relatives could be found during a study. The researchers believe that the chance that these things will happen is very small, but they cannot promise that you will avoid any risk.



## HOW WILL INFORMATION ABOUT ME BE KEPT PRIVATE?

Your privacy is very important to the researchers, and they will make every effort to protect it. Here are just a few of the steps they will take:

- 1) When your samples are sent to the researchers, no information identifying you (such as your name) will be sent. Samples will be identified by a unique code only.
- 2) The list that links the unique code to your name will be kept separate from your sample and health information. Any Biobank and SWOG staff with access to the list must sign an agreement to keep your identity confidential.
- Researchers that receive your sample and information from SWOG will not know who you are. Researchers must also sign an agreement that they will not try to find out who you are.
- 4) Information that identifies you will not be given to anyone, unless required by law.
- If research results are published, your name and other personal information will not be used.

# WHAT ARE THE POSSIBLE BENEFITS?

You will not benefit from taking part. Your samples may be helpful to research whether you do or do not have cancer.) The researchers, using the samples from you and others, might make discoveries that could help people in the future.

## ARE THERE ANY COSTS OR PAYMENTS?

There are no costs to you or your insurance. You will not be paid for taking part. If any of the research leads to new tests, drugs, or other commercial products, you will not share in any profits.

## WHAT IF I CHANGE MY MIND?

| If you decide you no longer want your samples to be used, you can call the study doctor, |
|---|
| , (insert name of study doctor for main trial) at |
| (insert telephone number of study doctor for main trial) who will |
| let the researchers know. Then, any samples that remain in the bank will no longer be used. |
| Samples or related information that have already been given to or used by researchers will not be |
| returned. |

If you decide to withdraw your specimens from a SWOG Specimen Repository in the future, a written withdrawal of consent should be submitted through your study doctor to the SWOG Operations Office. Please designate in the written withdrawal whether you would prefer to have the specimens destroyed or returned to the study doctor.



| WHAT | IF I | HAVE | <b>MORE</b> | <b>QUESTI</b> | ONS? |
|------|------|------|-------------|---------------|------|
| | | | | X | |

| If you have questions about the use of your samples for research, contact the study doctor, , (insert name of study doctor for main trial), at |
|---|
| (insert telephone number of study doctor for main trial). |
| Please circle your answer to show whether or not you would like to take part in each option (include only applicable questions): |
| SAMPLES FOR FUTURE RESEARCH STUDIES: |
| My samples and related information may be kept in a Biobank for use in future health research. |
| YES NO |
| This is the end of the section about optional studies. |
| My Signature Agreeing to Take Part in the Main Study |
| I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed copy of this form. I agree to take part in the main study and any additional studies where I circled 'yes'. |
| Participant's signature |
| Date of signature |



# Specimen Consent Supplemental Sheets

#### How are Specimens Used for Research?

#### Where do specimens come from?

A specimen may be from a blood sample or from bone marrow, skin, toenails or other body materials. People who are trained to handle specimens and protect donors' rights make sure that the highest standards of quality control are followed by SWOG. Your doctor does not work for SWOG, but has agreed to help collect specimens from many patients. Many doctors across the country are helping in the same way.

#### Why do people do research with specimens?

Research with specimens can help to find out more about what causes cancer, how to prevent it, how to treat it, and how to cure it. Research using specimens can also answer other health questions. Some of these include finding the causes of diabetes and heart disease, or finding genetic links to Alzheimer's.

#### What type of research will be done with my specimen?

Many different kinds of studies use specimens. Some researchers may develop new tests to find diseases. Others may develop new ways to treat or even cure diseases. In the future, some of the research may help to develop new products, such as tests and drugs. Some research looks at diseases that are passed on in families (called genetic research). Research done with your specimen may look for genetic causes and signs of disease.

#### How do researchers get the specimen?

Researchers from universities, hospitals, and other health organizations conduct research using specimens. They contact SWOG and request samples for their studies. SWOG reviews the way that these studies will be done, and decides if any of the samples can be used. SWOG gets the specimen and information about you from your hospital, and sends the specimen samples and some information about you to the researcher. SWOG will not send your name, address, phone number, social security number or any other identifying information to the researcher.

#### Will I find out the results of the research using my specimen?

You will not receive the results of research done with your specimen. This is because research can take a long time and must use specimen samples from many people before results are known. Results from research using your specimen may not be ready for many years and will not affect your care right now, but they may be helpful to people like you in the future.

#### Why do you need information from my health records?

In order to do research with your specimen, researchers may need to know some things about you. (For example: Are you male or female? What is your race or ethnic group? How old are you? Have you ever smoked?) This helps researchers answer questions about diseases. The information that will be given to the researcher may include your age, sex, race, diagnosis, treatments and family history. This information is collected by your hospital from your health record and sent to SWOG. If more information is needed, SWOG will send it to the researcher.

#### Will my name be attached to the records that are given to the researcher?

No. Your name, address, phone number and anything else that could identify you will be removed before they go to the researcher. The researcher will not know who you are.



#### How could the records be used in ways that might be harmful to me?

If your confidential genetic information is discovered, you may suffer from genetic discrimination. Genetic discrimination occurs if people are treated unfairly because of differences in their genes that increase their chances of getting a certain disease. In the past, this could have resulted in the loss of health insurance or employment. Because of this, The Genetic Information Nondiscrimination Act of 2008, also referred to as GINA, was passed by Congress to protect Americans from such discrimination. The new law prevents discrimination from health insurers and employers. This act was signed into federal law on May 21, 2008, and went into effect May 2009. This law does not cover life insurance, disability insurance and long-term care insurance.

While this study has safeguards in place to protect your confidential genetic information and to make it extremely unlikely that your identity would be connected with any special studies that are performed on your tissue, it is possible that this information could be discovered by someone who is unauthorized to have access to it.

#### How am I protected?

SWOG is in charge of making sure that information about you is kept private. SWOG will take careful steps to prevent misuse of records. Your name, address, phone number and any other identifying information will be taken off anything associated with your specimen before it is given to the researcher. This would make it very difficult for any research results to be linked to you or your family. Also, people outside the research process will not have access to results about any one person which will help to protect your privacy.

## What if I have more questions?

If you have any questions, please talk to your doctor or nurse, or call our research review board at (Insert IRB's Phone Number).

